CLINICAL TRIAL: NCT02948179
Title: Efficacy and Safety of Preimplantation Genetic Diagnosis in Blocking Pathogenic Gene Inheritance for Autosomal Dominant Polycystic Kidney Disease: a Multicenter Clinical Trial
Brief Title: Using Preimplantation Genetic Diagnosis in Autosomal Dominant Polycystic Kidney Disease Patients: a Multicenter Clinical Trial
Acronym: ESPERANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changlin Mei (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Shandong Provincial Hospital (Other Government); Tang-Du Hospital (Other); Shengjing Hospital (Other); Second Xiangya Hospital of Central South University (Other); Reproductive & Genetic Hospital of CITIC-Xiangya (Other); Peking University Third Hospital (Other); Navy General Hospital, Beijing (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The First Affiliated Hospital of Soochow University (Other); Sir Run Run Shaw Hospital (Other); Fuzhou General Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Wuhan TongJi Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Renmin Hospital of Wuhan University (Other); Xiangya Hospital of Central South University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Southwest Hospital, China (Other); LanZhou University (Other); Shaanxi Provincial People's Hospital (Other); West China Hospital (Other); West China Second University Hospital (Other); Sichuan Provincial People's Hospital (Other); Hebei Medical University Third Hospital (Other); Hebei Province Center for Reproductive Medicine (Unknown); The Second Hospital of Hebei Medical University (Other); Hospital for Reproductive Medicine Affiliated to Shandong University (Unknown)
Responsible Party: Sponsor-Investigator, Changlin Mei, Professor, Director of kidney Institute, Shanghai Changzheng Hospital
Organization: Shanghai Changzheng Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CZKIPLA-ADPKD-003
Record Dates: First submitted 2016-10-20; First posted 2016-10-28 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Polycystic Kidney, Type 1 Autosomal Dominant Disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preimplantation genetic diagnosis group (Experimental): ADPKD patients will complete the whole process of preimplantation genetic diagnosis with healthy baby without pathogenic gene inheritance.
  Interventions: Procedure: Preimplantation Genetic Diagnosis
- Natural pregnancy group (No Intervention): ADPKD patients, pathogenic mutations in PKD1, have natural pregnancy without preimplantation genetic diagnosis.The investigators will perform genetic tests on the blood or umbilical cord blood of infants born between January 2014 and June 2020.

INTERVENTIONS:
Procedure: Preimplantation Genetic Diagnosis — Using Preimplantation genetic diagnosis, including multiple annealing and looping-based amplification cycles amplification technique, the investigators have had screened out healthy embryos by In Vitro Fertilization. Then the investigators transplanted embryos returned to the parent. Finally, participants will have healthy baby without pathogenic gene inheritance.
  Arms: Preimplantation genetic diagnosis group

SUMMARY:
Autosomal dominant polycystic kidney disease (ADPKD) is the most common monogenic hereditary kidney disease in humans. ADPKD may affect all the generations of the ADPKD family and the probability of ADPKD is 50% in the second generation for each gender. It has been confirmed that PKD1 and PKD2 are two pathogenic genes of ADPKD. Nowadays, the investigators have established an effective gene detection technology platform for PKD1/2 gene with long fragment PCR and next generation sequencing. First, the investigators performed genetic testing in patients with clinically diagnosed ADPKD and strong fertility desire, but afraid of hereditary risk. Using Preimplantation genetic diagnosis, including multiple annealing and looping-based amplification cycles amplification technique, the investigators successfully screened out healthy embryos by In Vitro Fertilization. Then the investigators transplanted embryos returned to the parent. When the baby is born, using umbilical cord blood gene detection, the investigators confirmed that the neonates do not inherit genetic defects form parents. The investigators have succeeded in one couple. The investigators design a multicenter clinical trial to confirm those procedures efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Only one ADPKD patient in one couple without gender limitation
* Wife has age limitation from 20 years to 35 years
* ADPKD ADPKD diagnosis with or without family history
* Find out specific pathogenic mutations in the PKD1 gene with at least one of the following: one of family patients done kidney transplantation or renal replacement therapy before 58 years old; one of family patients died of complications before 55 years old; the patient with total kidney volume more than 650ml; the patient with total kidney volume increase rate more than 6% every year; the patient's PKD1 mutation belongs to truncated gene mutation.
* Both husband and wife have assisted reproductive conditions and will
* Pregnancy compliance with Chinese laws
* Signed informed consent

Exclusion Criteria:

* Active pathogenic microorganism infection, such as hepatitis B or C, HIV, pulmonary tuberculosis, giant cell virus, fungi or other contraindications for preimplantation genetic diagnosis and so on
* Any one of the couple has used any drugs which may lead to abnormal reproductive system function, reproductive cell abnormalities, pregnancy risk increases in the past 3 months, or has history of drug abuse
* Any one of the couple has malignancy
* The wife has uncontrolled hypertension or refractory hypertension
* The wife has diabetes mellitus
* The wife has albuminuria
* The wife has autoimmune disease
* The wife has other disorders or functional abnormalities, such as liver or renal dysfunction, which may be aggravated by pregnancy or assisted reproduction
* Allergy to drugs or related products which cannot avoid in our study
* Participating in other clinical studies in last 3 months
* Participants cannot follow the study program
* Other conditions that the researchers considered unsuitable for participation

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 459 (Actual)
Dates: Start 2016-09-02 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Healthy baby Rate without pathogenic gene inheritance | through study completion, an average of 2 year
  The investigators will do umbilical cord blood gene detection for the baby to confirm with or without pathogenic gene inheritance. The investigators will compare two groups of healthy newborns rate.

SECONDARY OUTCOMES:
Success rate in pretest of preimplantation genetic diagnosis | through study completion, an average of 2 year
  Using couples blood to do pretest of preimplantation genetic diagnosis in Peripheral blood mononuclear lymphocyte.
Technical failure rate of preimplantation genetic diagnosis. | Amniotic fluid puncture test (pregnancy 16 to 19 weeks ) and Birth day
  The rate of amniotic fluid puncture test or umbilical cord blood gene detection confirm the offspring containing pathogenic gene mutation.
Oocyte retrieval rate | through study completion, an average of 2 years
  The proportion of good eggs obtained after ovulation induction
Good quality embryo rate | through study completion, an average of 2 years
  The well-developed blastocyst ratio obtained after intracytoplasmic sperm injection
Pregnancy rate | Four weeks after embryo transplantation
  Successful pregnancy rate of transplanted embryo
Take home baby rate | Two week after neonatus birth day
  Healthy newborn birth rate in preimplantation genetic diagnosis group
The total kidney volume change rate | From enroll to postpartum 6 months
  The investigators do twice kidney MRI scan for calculating total kidney volume change rate between enroll and postpartum 6 months.
The estimated glomerular filtration rate change | From enroll to postpartum 6 months
  The investigators do twice serum creatinine test between enroll and postpartum 6 months, then using CKD-EPI formula to calculate eGFR.

OTHER OUTCOMES:
The incidence of ovarian hyperstimulation syndrome | through study completion, an average of 2 years
  the incidence of ovarian hyperstimulation syndrome
The incidence of organ injuries | through study completion, an average of 2 years
  the incidence of organ injuries
The incidence of infection | through study completion, an average of 2 years
  the incidence of infection
The incidence of abortion rate | through study completion, an average of 2 years
  the incidence of abortion rate

CONTACTS AND LOCATIONS:
Overall Officials: changlin Mei, Master, Principal Investigator — Institute of Nephrology, Changzheng Hospital; wen Li, doctor, Principal Investigator — Center of Reproductive Medicine, Changzheng Hospital
Locations (31):
- China (31):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Navy General Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Southwest Hospital, Chongqing, Chongqing Municipality
  - Fuzhou General Hospital, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Hebei Province Center for Reproductive Medicine, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Wuhan Tongji Hospital, Wuhan, Hubei
  - Wuhan Union Hospital, Wuhan, Hubei
  - Reproductive & Genetic Hospital of CITIC-Xiangya, Changsha, Hunan
  - Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Shengjing Hospital, Shenyang, Liaoning
  - Hospital for Reproductive Medicine Affiliated to Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Tang-Du Hospital, Xi’an, Shanxi
  - Shanxi Provincial People's Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - West China Second University Hospital, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No